CLINICAL TRIAL: NCT02988986
Title: Open Label, Phase II Trial of Neoadjuvant TAK-228 Plus Tamoxifen in Patients With Estrogen Receptor (ER)-Positive, Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Breast Cancer
Brief Title: TAK-228 Plus Tamoxifen in Patients With ER-Positive, HER2-negative Breast Cancer
Acronym: ANETT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jenny C. Chang, MD, Houston Methodist Cancer Center Director, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016065
Record Dates: First submitted 2016-11-30; First posted 2016-12-12 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Estrogen Receptor Positive Breast Cancer
Keywords: mTOR; Tamoxifen; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sapanisertib; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-228 Plus Tamoxifen (Experimental): TAK-228 will be orally administered at 30 mg weekly for 16 weeks.
  Tamoxifen will be orally administered at 20 mg daily for 16 weeks.
  Interventions: Drug: TAK-228; Drug: Tamoxifen

INTERVENTIONS:
Drug: TAK-228 — MTORC1/2 inhibitor
  Other Names: INK128, MLN0128
Drug: Tamoxifen — Non-steroidal anti-estrogen
  Other Names: Apo-Tamox, Gen-Tamoxifen, Nolvadex, Novo-Tamoxifen

SUMMARY:
This is an open label phase II clinical trial to determine the efficacy, toxicity, and safety of TAK-228 plus tamoxifen in patients with newly diagnosed ER-positive, HER2-negative breast cancer.

DETAILED DESCRIPTION:
The mTOR pathway is commonly dysregulated in ER-positive breast cancers and represents a key resistance mechanism to endocrine therapy such as tamoxifen. We plan to target the mTOR pathway with mTORC1/2 inhibitor TAK-228 to overcome tamoxifen resistance in early-stage ER-positive breast cancer. An open label phase II clinical trial will be conducted to determine the efficacy, toxicity, and safety of TAK-228 plus tamoxifen in patients with newly diagnosed ER-positive, HER2-negative breast cancer. TAK-228 (30 mg weekly) plus tamoxifen (20 mg daily) will be administered for 16 weeks. Patients will undergo tumor biopsy before starting the study treatment and after 6 weeks of study treatment. Blood samples for pharmacokinetics analysis will be obtained 1 hour before and after TAK-228 dosing on days 1 and 15 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male ≥ 18 years of age.
2. Newly diagnosed ER-positive, HER2-negative breast cancer. ER-positive is defined as ≥ 1% immunohistochemical (IHC) staining of any intensity. HER2 test result is negative if a single test (or both tests) performed show:

   * IHC 1+ or 0
   * In situ hybridization negative based on:

     * Single-probe average HER2 copy number < 4.0 signals/cell
     * Dual-probe HER2/CEP17 ratio < 2 with an average HER2 copy number < 4.0 signals/cell.
3. Patients with stage II-III breast cancer are eligible if they are deemed appropriate for neoadjuvant endocrine therapy by the referring or treating medical oncologist. Patients with stage I disease are eligible if they are deemed borderline candidates for breast conservation and the treating surgeon recommends preoperative therapy to increase the chances of breast conservation.
4. Eastern Cooperative Oncology Group performance status and/or other performance status of ≤ 1.
5. Female patients who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 effective method of contraception and 1 additional effective (barrier) method, at the same time, from the time of signing the ICF through 90 days (or longer, as mandated by local labeling [e.g., United Surgical Partners International, summary of product characteristics, etc.] after the last dose of the study drugs, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient (periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condom should not be used together).
6. Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

   * Agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of the study drugs, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient
   * Agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of the study drugs.
7. Screening clinical laboratory values as specified below:

   1. Bone marrow reserve consistent with: absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL (without transfusion) within 1 week preceding the administration of the study drugs;
   2. Hepatic status: Serum total bilirubin ≤ 1 x upper limit of normal (ULN; in the case of known Gilbert's syndrome, a higher serum total bilirubin [< 1.5 x ULN] is allowed), aspartate aminotransferase and alanine aminotransferase ≤ 1.5 x ULN, and alkaline phosphatase ≤ 1.5 x ULN;
   3. Renal status: Creatinine clearance ≥50 mL/min based on Cockcroft-Gault estimate or based on urine collection (12 or 24 hour);
   4. Metabolic status: HbA1c < 7.0%, fasting serum glucose ≤ 130 mg/dL, and fasting triglycerides ≤ 300 mg/dL.
8. Ability to swallow oral medications.
9. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
10. Negative serum pregnancy test within 7 days prior to the administration of the study drugs for female patients of childbearing potential.
11. Patient must be accessible for treatment and follow-up.
12. Patient must be willing to undergo breast biopsies as required by the study protocol.

Exclusion Criteria:

1. Any patient with metastatic disease.
2. Other clinically significant comorbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise the patient's participation in the study.
3. Known human immunodeficiency virus infection.
4. Known hepatitis B surface antigen-positive or known or suspected active hepatitis C infection.
5. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of the protocol-specified treatment.
6. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of the study drugs or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
7. Breastfeeding or pregnant.
8. Manifestations of malabsorption due to prior gastrointestinal surgery, gastrointestinal disease, or an unknown reason that may alter the absorption of TAK-228. Patients with enteric stomata are also excluded.
9. Treatment with any investigational products within 2 weeks before administration of the first dose of the study drugs.
10. Poorly controlled diabetes mellitus (defined as HbA1c > 7%). Patients with a history of transient glucose intolerance due to corticosteroid administration may be enrolled in the study if all other inclusion criteria and none of the other exclusion criteria are met.
11. History of any of the following within the last 6 months before administration of the first dose of the study drugs:

    * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
    * Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures
    * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation, and ventricular tachycardia)
    * Placement of a pacemaker for control of rhythm
    * New York Heart Association Class III or IV heart failure
    * Pulmonary embolism
12. Significant active cardiovascular or pulmonary disease including:

    * Uncontrolled hypertension (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg). Use of antihypertensive agents to control hypertension before week 1, day 1 is allowed.
    * Pulmonary hypertension
    * Uncontrolled asthma or O2 saturation < 90% by arterial blood gas analysis or pulse oximetry on room air
    * Significant valvular disease, severe regurgitation, or stenosis by imaging independent of symptom control with medical intervention or history of valve replacement
    * Medically significant (symptomatic) bradycardia
    * History of arrhythmia requiring an implantable cardiac defibrillator
    * Baseline QTc prolongation (e.g., repeated demonstration of QTc interval > 480 milliseconds or history of congenital long QT syndrome or torsades de pointes)
13. Treatment with strong inhibitors and/or inducers of CYP3A4, CYP2C9, or CYP2C19 within 7 days preceding the first dose of the study drugs.
14. Patients receiving systemic corticosteroids (either IV or oral steroids, excluding inhalers or low-dose hormone replacement therapy) within 1 week before administration of the first dose of the study drugs.
15. Daily or chronic use of a proton pump inhibitor (PPI) and/or having taken a PPI within 7 days before receiving the first dose of the study drugs.
16. Patients unwilling or unable to comply with the study protocol.
17. Patients previously treated with hormonal therapy (tamoxifen, AI) or PI3K, AKT, dual PI3K/mTOR, TORC1/2, or mTORC1 inhibitors.
18. Patients who are currently being treated with cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) other than the trial therapy.
19. Patients with hypersensitivity to mTOR inhibitors or tamoxifen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny C Chang, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (3):
- United States (3):
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Hospital Willowbrook, Houston, Texas
  - Houston Methodist Hospital Sugar Land, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data and materials on human subjects will be shared with other eligible investigators through appropriate means in accordance with the NIH policy on Sharing Research Data (NIH Guide, February 26, 2003). Data will be also shared with the funding agency and regulatory agencies as required. Data will be shared with other investigators within the limits of HIPAA and other patient confidentiality requirements. This will generally require removal of all patient identifiers for all source documents and the use of arbitrarily assigned one-way identifiers. In some cases, requestors will be asked to sign a formal data sharing agreement that will provide for a commitment to use data only for research purposes and not to identify individuals, keep the data secure, and destroy or return data after analyses are complete. Prior approval will be obtained from collaborating investigators, research sponsors, and/or other stake-holders before sharing if proprietary information or products are involved.
Time Frame: From study end (3/30/2019) for 5 years.
Access Criteria: Data and materials on human subjects will be shared with other eligible investigators through appropriate means in accordance with the NIH policy on Sharing Research Data (NIH Guide, February 26, 2003). Data will be also shared with the funding agency and regulatory agencies as required. Data will be shared with other investigators within the limits of HIPAA and other patient confidentiality requirements. This will generally require removal of all patient identifiers for all source documents and the use of arbitrarily assigned one-way identifiers. In some cases, requestors will be asked to sign a formal data sharing agreement that will provide for a commitment to use data only for research purposes and not to identify individuals, keep the data secure, and destroy or return data after analyses are complete. Prior approval will be obtained from collaborating investigators, research sponsors, and/or other stake-holders before sharing if proprietary information or products are involved.

RESULTS

PARTICIPANT FLOW:
Groups:
- TAK-228 Plus Tamoxifen: TAK-228 will be orally administered at 30 mg weekly for 16 weeks.
  Tamoxifen will be orally administered at 20 mg daily for 16 weeks.
  TAK-228: MTORC1/2 inhibitor
  Tamoxifen: Non-steroidal anti-estrogen
Period: Overall Study
Arm/Group | TAK-228 Plus Tamoxifen
Started | 28
Completed | 25
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | TAK-228 Plus Tamoxifen
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Twenty-eight women were enrolled on the trial, and 25 completed the entire study course. Population: 28 patients were enrolled in the study. 25 completed the entire study. 23 were evaluable for the primary endpoint. All 28 patients were evaluated for safety and toxicity.
  years | 52 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
Stage I-III ER-positive, HER-2 negative breast cancer [Count of Participants; unit: Participants] | 28

OUTCOME MEASURES:

1. Primary Outcome: Ki67 Expression
Description: Ki67 expression change from baseline to 6 weeks
Time Frame: Baseline to 6 weeks
Population: Change in baseline Ki67 expression at 6 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of cells with Ki67 expression
Arm/Group | TAK-228 Plus Tamoxifen
Number analyzed (Participants) | 23
Percentage of cells with Ki67 expression
  Ki67 expression at baseline | 15 [10 to 25]
  Ki67 expression at 6 weeks | 10 [2 to 38]
Statistical Analysis 1: Comparison: TAK-228 Plus Tamoxifen; The primary endpoint was the change in Ki67 after 6 weeks of treatment; Test type: Superiority — Based on prior data for Ki67 changes in the tamoxifen arm alone, we will assume null hypothesis and alternative hypotheses of 60% and 80% reduction in Ki67, respectively. A sample of 25 patients will provide 86% power to detect the hypothesized reduction in Ki67 with 5% alpha based on a two-sided, one sample t-test of mean percent change in Ki67 level; p = 0.0023, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants Meeting Certain Preoperative Endocrine Prognostic Index (PEPI)
Description: Evaluate the number of participants meeting certain PEPI score after treatment with TAK-228 plus tamoxifen.
  PEPI score of 0 indicates low risk of disease recurrence (better outcome) PEPI score of 1-3 indicates intermediate risk of of disease recurrence (worse outcome) PEPI score of >4 indicates high risk of of disease recurrence (worst outcome)
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Tamoxifen: 20 mg p.o QW x16 weeks
Arm/Group | Tamoxifen
Number analyzed (Participants) | 21
Participants
  PEPI score of 0 | 0
  PEPI score of 1-3 | 6
  PEPI score of >4 | 15

3. Secondary Outcome: Number of Participants With Pathological Complete Response (pCR)
Description: Pathologic complete response was defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0 ypN0 or ypTis ypN0 in the current American Joint Committee on Cancer staging system).
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-228 Plus Tamoxifen
Number analyzed (Participants) | 23
Participants | 0

4. Other Pre Specified Outcome: Plasma Concentrations of TAK-228 Plus Tamoxifen
Description: Measure plasma concentrations of TAK-228 plus tamoxifen over time
Time Frame: 16 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Correlation Between Change in Ki67 Expression and pCR to TAK-228 Plus Tamoxifen
Description: Assess the correlation between change in Ki67 expression and pCR to TAK-228 plus tamoxifen
Time Frame: 16 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Correlation Between Tumor Mutational Status and Response to TAK-228 Plus Tamoxifen
Description: Assess correlation between tumor mutational status and response to TAK-228 plus tamoxifen
Time Frame: 16 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Correlation Between Change in mTOR Expression and pCR to TAK-228 Plus Tamoxifen
Description: Assess the correlation between change in mTOR expression and pCR to TAK-228 plus tamoxifen
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Groups:
- TAK-228 and Tamoxifen: 20 mg p.o QW x16 weeks
Arm/Group | TAK-228 and Tamoxifen
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-228 and Tamoxifen (N=28)
hyperglycemia (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-228 and Tamoxifen (N=28)
Nausea (Gastrointestinal disorders) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT02988986/Prot_SAP_002.pdf